CLINICAL TRIAL: NCT00735332
Title: A Phase IIa Study of TLN-232 as Second-line Therapy for Patients With Metastatic Melanoma
Brief Title: Efficacy Study of TLN-232 in Patients With Recurring Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: License termination.
Sponsor: Thallion Pharmaceuticals (Industry)
Responsible Party: Didier Reymond, MD / Executive Vice-President Clinical Development, Thallion Pharmaceuticals Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLN-232-202
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma; Phase II; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm (Experimental)
  Interventions: Drug: TLN-232

INTERVENTIONS:
Drug: TLN-232 — 21 day continuous IV administration of TLN-232 followed by a 7-day recovery period
  Other Names: Formerly CAP-232

SUMMARY:
The objective of this study is to assess the efficacy and safety of TLN-232 used to treat patients with metastatic melanoma that recur/progress after receiving first line systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV (M1a, M1b, and M1c) unresectable metastatic melanoma (cutaneous, mucosal or acral lentiginous)
* First progression after treatment by one first line systemic therapy for metastatic melanoma (immunotherapy or targeted therapy or chemotherapy or any combination of them)
* Measurable recurrent/progressive disease by radiological scan ≤ 21 days prior to Day 1, Cycle 1
* Age ≥ 18 years
* ECOG ≤ 2
* Normal organ and marrow function as defined below:

  * Leukocytes ≥2.5 x 109/L
  * Absolute neutrophil count ≥1.5 x 109/L
  * Platelets ≥100 x 109/L
  * Hemoglobin ≥100 g/L (10g/dL)
  * Total bilirubin ≤1.5 X institutional ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional ULN
  * Creatinine ≤1.5 X institutional ULN

Exclusion Criteria:

* Patients with a life expectancy ≤ 16 weeks
* Patients with ocular melanoma
* Patients with symptomatic and/or unstable brain metastasis during the last 3 months (90 days) prior to Day 1, Cycle 1
* Patients with a history of allergic reactions or hypersensitivity to somatostatin analogues
* Patients with a documented history of HIV, active hepatitis B or C infection
* Female patients who are pregnant or lactating
* Patients who are receiving hormonal therapy (with the exception of hormone replacement therapy and hormonal contraceptives), systemic steroids, immunosuppressive therapy or coumadin (low molecular weight heparin is permitted)
* Patients with grade ≥2 peripheral neuropathy (CTCAE criteria)
* Patients in whom a proper central line cannot be established

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of TLN-232 in patients with recurrent metastatic melanoma measured by overall response rate at 16 weeks from date of initial infusion of TLN-232 (Day 1, Cycle 1). | Complete response, partial response or stable disease at 16 weeks from date of initial infusion of TLN-232 (Day 1, Cycle 1)

SECONDARY OUTCOMES:
To examine the safety and tolerability of TLN-232 in patients with recurrent metastatic melanoma | Maximum 13 months from date of initial infusion of TLN-232 (Day 1, Cycle 1)

CONTACTS AND LOCATIONS:
Overall Officials: David Hogg, MD, Principal Investigator — Princess Margaret Hospital, Toronto
Locations (4):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Notre-Dame du CHUM, Montreal, Quebec